CLINICAL TRIAL: NCT01309412
Title: A Phase 1 Study of CNTO 328 (Siltuximab) in Combination With Bortezomib and Dexamethasone for Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Phase 1 Study of CNTO 328 (Siltuximab) in Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Protocol was stopped due to the safety issue in Global
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017737; JPN-C0328-MM-101 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or refractory multiple myeloma; CNTO 328; siltuximab; bortezomib; dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Siltuximab (Experimental): Siltuximab 5.5 or 11.0 mg/kg by intravenous infusion over 1 hour on Day 1 of each 21-day cycle until progression
  Interventions: Drug: Siltuximab

INTERVENTIONS:
Drug: Siltuximab — 5.5 or 11.0 mg/kg by intravenous infusion over 1 hour on Day 1 of each 21-day cycle until progression

SUMMARY:
The purpose of this study is to assess the safety and the tolerability of siltuximab up to 11.0 mg/kg in combination with bortezomib and dexamethasone for patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This study is an open-label (both physician and patient know the name of the study drug), multicenter (more than one site) study of siltuximab in patients with relapsed or refractory multiple myeloma receiving siltuximab in combination with bortezomib/dexamethasone to evaluate the safety, pharmacokinetics (how drugs are absorbed in the body, how they are distributed within the body and how they are removed from the body over time), efficacy and immunogenicity (the ability to induce immune responses). This study is planned with a dose escalation of siltuximab to levels of 5.5 mg/kg (Dose Level 1) and 11.0 mg/kg (Dose Level 2) given intravenously. Recommended doses will be determined based on the incidence of dose-limiting toxicity in patients with relapsed or refractory multiple myeloma when siltuximab at dose levels of 5.5 mg/kg and 11.0 mg/kg is administered with bortezomib/dexamethasone. Treatment with siltuximab will be started at Dose Level 1, and treatment at Dose Level 2 will not be started until completing the safety evaluation at the end of the observation period of Cycle 1 for all patients at Dose level 1. Once 11.0 mg/kg is determined as a recommended dose, the dose for patients whose starting dose is 5.5 mg/kg, and who have not achieved complete response, can be escalated to 11.0 mg/kg based on patient consent and investigator discretion in the next cycle. Siltuximab will be given at 5.5 or 11.0 mg/kg by intravenous infusion over 1 hour on Day 1 of each 21-day cycle until progression. Twice-weekly intravenous administration of bortezomib 1.3 mg/m2 (Days 1, 4, 8, and 11) will be followed by a 10-day rest period (Days 12-21). Four-per-week oral administration of dexamethasone 20 mg (Days 1, 2, 4, 5, 8, 9, 11 and 12) will be followed by a 9-day rest period (Days 13-21).

ELIGIBILITY:
Inclusion Criteria:

* Patients proven to have symptomatic or nonsecretory multiple myeloma
* Patients with a measurable lesion
* Patients who have previously received 1-3 regimens for multiple myeloma
* Patients must have progressed on or be refractory to the most recent line of treatment
* Patients with Eastern Cooperative Oncology Group performance status of 0-2
* Patients having the following laboratory values within 14 days before the scheduled day of initial administration of the study drug: hemoglobin 8 g/dL or more, absolute neutrophil count 1,000/mm3 or more, platelet count 50,000/mm3 or more, aspartate aminotransferase, and alanine aminotransferase 2.5 times or more of upper limit of normal range, total bilirubin 1.5 times or more of upper limit of normal range, calculated creatinine clearance 20 mL/min or more, corrected serum calcium less than 12.5 mg/dL

Exclusion Criteria:

* Patients with primary amyloidosis, plasma cell leukemia or other conditions in which M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Patients with Grade 1 peripheral neuropathy with pain or Grade 2 or higher peripheral neuropathy
* Patients who have undergone allogeneic bone marrow transplantation within 28 days before the start of treatment with the study drug
* Patients who have been exposed to agents targeting interleukin-6 (IL-6) or the IL-6 receptor
* Patients refractory to bortezomib
* Patients having treatment discontinued because of the toxicity of bortezomib
* Patients requiring dose reduction because of the toxicity of bortezomib
* Patients who have received chemotherapy, plasmapheresis or radiation therapy within 21 days before the start of treatment (within 42 days for nitrosoureas)
* Patients who have undergone major surgery including open biopsy (excluding bone marrow) within 21 days before study treatment or planning to have surgery (except for minor surgical procedures) during the study
* Human immunodeficiency virus antibody-positive, hepatitis C virus antibody-positive or hepatitis B surface antigen-positive patients
* Patients with known hypersensitivity to boron or mannitol
* Patients with a history of unmanageable severe infusion reactions to monoclonal antibodies or to murine, chimeric or human proteins or their excipients
* Patients with concurrent medical condition that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in the study
* Patients with significant cardiac disease characterized by significant ischemic coronary disease, significant arrhythmias, or congestive heart failure (New York Heart Association Class III or IV) or myocardial infarction within 6 months before the first dose of study drug
* Patients who are clinically diagnosed with pneumonitis (interstitial pneumonia) or pulmonary fibrosis or have abnormal interstitial shadows bilaterally on chest CT, with or without symptoms

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events as a measure of safety and tolerability | Up to 14 months

SECONDARY OUTCOMES:
Serum siltuximab concentration | Maximum 15 weeks
Number of patients with a positive immune response to siltuximab | Up to 14 months
Number of patients with an overall response (complete response and partial response) | Up to 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (5):
- Japan (5):
  - Isehara
  - Kyoto
  - Nagoya
  - Niigata
  - Tokyo

REFERENCES:
- [Derived] Suzuki K, Ogura M, Abe Y, Suzuki T, Tobinai K, Ando K, Taniwaki M, Maruyama D, Kojima M, Kuroda J, Achira M, Iizuka K. Phase 1 study in Japan of siltuximab, an anti-IL-6 monoclonal antibody, in relapsed/refractory multiple myeloma. Int J Hematol. 2015 Mar;101(3):286-94. doi: 10.1007/s12185-015-1743-y. Epub 2015 Feb 6. PMID 25655379
- See also: A Phase 1 Study of CNTO 328 (siltuximab) in Combination with Bortezomib and Dexamethasone for Subjects with Relapsed or Refractory Multiple Myeloma — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=443&filename=CR107737_CSR.pdf